CLINICAL TRIAL: NCT01914978
Title: Living Confidently With Food Allergy: Evaluating the Effectiveness of a Handbook for the Newly Diagnosed
Brief Title: Evaluating the Effectiveness of a Handbook for Parents of Children Newly Diagnosed With Food Allergy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Jennifer LeBovidge, Psychologist, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-P00007167
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Hypersensitivity, Food
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Handbook (Experimental): Food allergy handbook for parents
  Interventions: Other: Food allergy handbook for parents
- Treatment as usual (Placebo Comparator): Food allergy treatment as usual
  Interventions: Other: Food allergy treatment as usual

INTERVENTIONS:
Other: Food allergy handbook for parents — The food allergy handbook was designed to be a reliable resource to supplement physician management of food allergy, addressing key topics central to effective allergy management and maintenance of positive quality of life. The handbook includes evidence-based information about food allergies and their management, practical strategies for transferring allergy management skills into daily life, strategies for educating others about allergies, strategies for coping with common emotional challenges associated with food allergy, and strategies for teaching children and involving them in allergy management.
  Arms: Handbook
Other: Food allergy treatment as usual
  Arms: Treatment as usual

SUMMARY:
The objective of this research is to evaluate the effectiveness of a handbook for parents of children newly diagnosed with food allergy. The handbook was developed to provide information and strategies to support families in effectively managing food allergies while maintaining positive quality of life. Parents of children newly diagnosed with food allergy (within the past year) will be randomized into either the treatment condition (handbook) or a control condition (management of food allergy as usual). Participants will complete study questionnaires online at three time points: baseline (this will be before receiving the handbook for the treatment group), post-intervention (2-3 weeks after baseline), and follow-up (2-3 months after baseline). Data will be analyzed for change on study outcome measures and satisfaction with the handbook. Parents in the control group will receive the handbook following the conclusion of their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children ages 0 to 18 years newly diagnosed with food allergy (within the past 12 months)
* Child's food allergy has been diagnosed by a physician
* Child has been prescribed an epinephrine auto-injector

Exclusion Criteria:

* Non-English speakers, as the handbook (study intervention) is only available in English at this time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in food allergy-specific quality of life score | 2 week and 2-month follow-up
  Food Allergy-specific quality of life measured on the Food Allergy Quality of Life-Parental Burden Questionnaire (total score)

SECONDARY OUTCOMES:
Changes in food allergy knowledge score | 2-week and 2-month follow-up
  Food allergy knowledge questions will include a subset of questions from the Chicago Food Allergy Research Survey for Parents of Children with Food Allergy (CFAR-PRNT) and questions developed by the investigators
Change in confidence in allergy management skills score | 2-week and 2-month follow-up
  This questionnaire was developed for the current study, to assess parent's level of confidence in various allergy management skills (e.g., understanding food labels, knowing the symptoms of an allergic reaction, teaching babysitters, relatives and other caregivers how to take care of your child's allergies, etc)
Change in food allergy outcome expectations score | 2-week and 2-month follow-up
  The Food Allergy Independent Measure (FAIM) consists of four questions assessing the parents' expectations of outcomes related to a child's food allergy (i.e., likelihood of the child accidentally ingesting an allergenic food, experiencing a severe reaction, dying following accidental ingestion, and receiving effective treatment in the event of accidental ingestion), which have been associated with health-related quality of life associated with food allergy.
Parent satisfaction with study handbook (study intervention) | 2-week follow-up
  Defined by at least 80% of parents indicating positive ratings of usefulness, novelty of content, clarity of content, and [lack of] distress associated with content, [lack of] distress associated with content, and [lack of] barriers to use of the handbook.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S LeBovidge, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] LeBovidge JS, Michaud A, Deleon A, Harada L, Waserman S, Schneider L. Evaluating a handbook for parents of children with food allergy: a randomized clinical trial. Ann Allergy Asthma Immunol. 2016 Mar;116(3):230-236.e1. doi: 10.1016/j.anai.2016.01.001. Epub 2016 Feb 3. PMID 26851890